CLINICAL TRIAL: NCT00394901
Title: A 13-Week, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study To Evaluate Efficacy And Safety Of Pregabalin In The Treatment Of Postherpetic Neuralgia
Brief Title: A 13-Week, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study Of Pregabalin For Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081120
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2009-02-27 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2010-02

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pregabalin 150mg/day (Experimental)
  Interventions: Drug: Pregabalin
- Pregabalin 300mg/day (Experimental)
  Interventions: Drug: Pregabalin
- Pregabalin 600mg/day (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo — placebo, oral administration for 13 weeks (1 week titration and 12-week fixed dose).
  Arms: Placebo
Drug: Pregabalin — Pregabalin 150mg/day (75mg BID), oral administration for 13 weeks (1-week titration and 12-week fixed dose).
  Arms: Pregabalin 150mg/day
Drug: Pregabalin — Pregabalin 300mg/day (150mg/BID), oral administration for 13 weeks (1-week titration and 12-week fixed dose).
  Arms: Pregabalin 300mg/day
Drug: Pregabalin — Pregabalin 600 mg/day (300 mg/BID), oral administration for 13 weeks (1-week titration and 12-week fixed dose).
  Arms: Pregabalin 600mg/day

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of pregabalin in the treatment of postherpetic neuralgia in a dose-ranging manner.

ELIGIBILITY:
Inclusion Criteria:

* Visual Analogue Scale (VAS) of pain is higher than 40 mm.
* Pain is sustained for more than 3 months after healing of herpes zoster skin rash.

Exclusion Criteria:

* Malignancy within the past 2 years.
* Patients who have undergone neurolytic or neurosurgical therapy for postherpetic neuralgia.
* Creatinine clearance </= 30 mL/min (estimated from serum creatinine, body weight, age, and sex using the Cockcroft and Gault equation, by omitting any decimal fractions).
* Patients having other severe pain which may impair the self assessment of the pain due to postherpetic neuralgia.
* Skin conditions in the affected dermatome that could alter sensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- Japan (39):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Ichikawa, Chiba
  - Pfizer Investigational Site, Urayasu, Chiba
  - Pfizer Investigational Site, Kasuga, Fukuoka
  - Pfizer Investigational Site, Kasuya-gun, Fukuoka
  - Pfizer Investigational Site, Maebaru-chūō, Fukuoka
  - Pfizer Investigational Site, Maebashi, Gunma
  - Pfizer Investigational Site, Takasaki, Gunma
  - Pfizer Investigational Site, Asahikawa, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Akashi, Hyōgo
  - Pfizer Investigational Site, Amagasaki, Hyōgo
  - Pfizer Investigational Site, Himeji, Hyōgo
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Nishinomiya, Hyōgo
  - Pfizer Investigational Site, Tsuchiura, Ibaraki
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Beppu, Ohita
  - Pfizer Investigational Site, Kishiwada, Osaka
  - Pfizer Investigational Site, Takatsuki, Osaka
  - Pfizer Investigational Site, Kawaguchi, Saitama
  - Pfizer Investigational Site, Kitamoto, Saitama
  - Pfizer Investigational Site, Tokorozawa, Saitama
  - Pfizer Investigational Site, Adachi-ku, Tokyo
  - Pfizer Investigational Site, Arakawa-ku, Tokyo
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Mitaka, Tokyo
  - Pfizer Investigational Site, Nakano-ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Suginami-ku, Tokyo
  - Pfizer Investigational Site, Toshima-ku, Tokyo
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Fukushima
  - Pfizer Investigational Site, Osaka
  - Pfizer Investigational Site, Saitama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081120&StudyName=A%2013-Week%2C%20Randomized%2C%20Double-Blind%2C%20Multicenter%2C%20Placebo-Controlled%20Study%20Of%20Pregabalin%20For%20Postherpetic%20Neuralgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty (50) centers in Japan
Pre-assignment Details: After a 1-week baseline phase, subjects were stratified into 1 of 2 strata based on their creatinine clearance (CLcr) values (Low, 30 <CLcr <=60 mL/min or Normal, CLcr > 60 mL/min) and then equally randomized into 1 of 4 treatment groups.
Groups:
- Placebo: During a 13-week double-blind phase, subjects received matching placebo.
- Pregabalin 150 mg/Day: During a 13-week double-blind phase, subjects received pregabalin 150 mg/day.
- Pregabalin 300 mg/Day: During a 13-week double-blind phase, after 1 week of up titration, subjects received pregabalin 300 mg/day for 12 weeks.
- Pregabalin 600 mg/Day: During a 13-week double-blind phase, after 1 week of up titration, subjects with low CLcr received pregabalin 300 mg/day and subjects with normal CLcr received pregabalin 600 mg/day for 12 weeks.
Period: Baseline Phase
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Started | 98 (Subjects randomized) | 87 (Subjects randomized) | 90 (Subjects randomized) | 97 (Subjects randomized)
Completed | 98 | 87 | 89 | 97
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Period: Double-blind Phase
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Started | 98 (Subjects treated with the study drug.) | 87 (Subjects treated with the study drug.) | 89 (Subjects treated with the study drug.) | 97 (Subjects treated with the study drug.)
Completed | 83 | 73 | 71 | 70
Not Completed | 15 | 14 | 18 | 27
Not completed — Adverse Event | 5 | 7 | 16 | 20
Not completed — Lack of Efficacy | 6 | 4 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Subject's Personal Reason | 1 | 0 | 0 | 1
Not completed — Lack of Compliance | 0 | 3 | 0 | 0
Not completed — Entry into another study was found | 0 | 0 | 1 | 0
Not completed — Found not to meet entrance criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day | Total
Number analyzed (Participants) | 98 | 87 | 89 | 97 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.6) | 70.2 (9.2) | 70.9 (9.8) | 68.4 (12.5) | 70.1 (10.2)
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 44 years | 2 | 1 | 2 | 6 | 11
  Between 45 and 64 years | 12 | 17 | 15 | 20 | 64
  >=65 years | 84 | 69 | 72 | 71 | 296
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 44 | 44 | 44 | 173
  Male | 57 | 43 | 45 | 53 | 198
Region of Enrollment [Number; unit: participants]
  Japan | 98 | 87 | 89 | 97 | 371

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Scores at Endpoint
Description: Endpoint mean pain score is defined as the mean of the last 7 daily pain diary rating while taking the study medication, up to and including day after last dose. Scores range from 0-10 (11 points ordinal) with higher scores indicating increased pain.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
score on scale | 5.12 (0.19) | 4.81 (0.20) | 4.26 (0.20) | 4.49 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.262, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.31, 95% CI [-0.85 to 0.23]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.002, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.86, 95% CI [-1.39 to -0.32]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.019, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.63, 95% CI [-1.15 to -0.10]

2. Primary Outcome: Mean Pain Score at Endpoint by Groups of Subjects With Expected Similar Plasma Concentrations
Description: as for outcome 1
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Groups:
- Placebo: Subjects who received matching placebo during a 13-week double-blind treatment phase.
- Expected Pregabalin Exposure of 300 mg/Day: Subjects with low CLcr (> 30 and <= 60 mL/min) who received pregabalin 150 mg/day and subjects with normal CLcr (> 60 mL/min) who received pregabalin 300 mg/day.
- Expected Pregabalin Exposure of 600 mg/Day: Subjects with low CLcr (> 30 and <= 60 mL/min) who received pregabalin 300 mg/day and subjects who received pregabalin 600 mg/day.
Arm/Group | Placebo | Expected Pregabalin Exposure of 300 mg/Day | Expected Pregabalin Exposure of 600 mg/Day
Number analyzed (Participants) | 97 | 92 | 122
score on scale | 4.99 (0.18) | 4.35 (0.19) | 4.34 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Expected Pregabalin Exposure of 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.016, ANCOVA; The model included treatment group modified based on the expected pregabalin exposure as a factor, and baseline score as covariate; Mean Difference (Final Values) = -0.64, 95% CI [-1.16 to -0.12]
Statistical Analysis 2: Comparison: Placebo vs Expected Pregabalin Exposure of 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.008, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.66, 95% CI [-1.14 to -0.17]

3. Primary Outcome: Number of Responders
Description: A responder is defined as a subject with a 50% reduction in weekly mean pain score from baseline to endpoint.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
participants | 15 | 21 | 32 | 30
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Proportion of responders were used for the statistical analyses. Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.1160, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0107, Cochran-Mantel-Haenszel; stratified by CLcr stratum

4. Primary Outcome: Mean Pain Scores at Week 1
Description: Weekly mean pain score is defined as the mean of the last 7 daily diary pain ratings. Scores range from 0-10 (11 points ordinal)with higher scores indicating increased pain.
Time Frame: Week 1
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
score on scale | 5.96 (0.17) | 5.45 (0.18) | 5.21 (0.18) | 5.23 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.038, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.51, 95% CI [-0.99 to -0.03]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.002, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.75, 95% CI [-1.22 to -0.27]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.002, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.72, 95% CI [-1.19 to -0.26]

5. Primary Outcome: Mean Pain Scores at Week 2
Description: as for outcome 4
Time Frame: Week 2
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 96 | 83 | 83 | 86
score on scale | 5.75 (0.17) | 5.27 (0.18) | 4.76 (0.18) | 4.73 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.048, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.48, 95% CI [-0.97 to 0.00]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.99, 95% CI [-1.47 to -0.52]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.03, 95% CI [-1.49 to -0.56]

6. Primary Outcome: Mean Pain Scores at Week 3
Description: as for outcome 4
Time Frame: Week 3
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 92 | 83 | 80 | 84
score on scale | 5.59 (0.17) | 5.18 (0.18) | 4.63 (0.18) | 4.60 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.096, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.41, 95% CI [-0.89 to 0.07]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.96, 95% CI [-1.44 to -0.48]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.99, 95% CI [-1.46 to -0.52]

7. Secondary Outcome: Endpoint Sensory Scores of the Short-Form McGill Pain Questionnaire
Description: Sensory score range from 0-33. Higher scores indicate more severe pain.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
score on scale | 8.97 (0.57) | 8.42 (0.61) | 7.11 (0.60) | 6.97 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.505, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.55, 95% CI [-2.16 to 1.06]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.023, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.86, 95% CI [-3.46 to -0.26]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.012, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.00, 95% CI [-3.56 to -0.44]

8. Secondary Outcome: Endpoint Affective Scores of the Short-Form McGill Pain Questionnaire
Description: Affective score range from 0-12. Higher scores indicate more severe pain.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 88 | 97
score on scale | 2.43 (0.22) | 2.14 (0.23) | 1.72 (0.23) | 1.82 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.349, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.29, 95% CI [-0.91 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.024, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.71, 95% CI [-1.32 to -0.10]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.045, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.61, 95% CI [-1.21 to -0.01]

9. Secondary Outcome: Endpoint Total Scores of the Short-Form McGill Pain Questionnaire
Description: Total score range from 0-45. Higher scores indicate more severe pain.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
score on scale | 11.39 (0.75) | 10.56 (0.79) | 8.84 (0.79) | 8.78 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.441, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.83, 95% CI [-2.93 to 1.28]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.017, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.55, 95% CI [-4.64 to -0.46]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.012, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.61, 95% CI [-4.65 to -0.56]

10. Secondary Outcome: Endpoint Visual Analogue Scale Scores of the Short-Form McGill Pain Questionnaire
Description: Visual Analogue Scale Score range from 0-100mm. Higher scores indicate more severe pain.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
mm | 50.02 (2.15) | 47.80 (2.28) | 41.99 (2.25) | 42.59 (2.14)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.470, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.23, 95% CI [-8.28 to 3.83]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.008, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -8.04, 95% CI [-14.0 to -2.06]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.013, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -7.43, 95% CI [-13.3 to -1.59]

11. Secondary Outcome: Endpoint Present Pain Intensity Scores of the Short-Form McGill Pain Questionnaire
Description: Present pain intensity score range from 0-5. Higher scores indicate more severe pain.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 96
score on scale | 2.21 (0.10) | 2.01 (0.11) | 1.78 (0.11) | 1.90 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.178, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.20, 95% CI [-0.48 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.003, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.43, 95% CI [-0.72 to -0.15]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.030, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.31, 95% CI [-0.59 to -0.03]

12. Secondary Outcome: Mean Sleep Interference Scores at Endpoint
Description: Scores range from 0-10. Higher scores indicate more severe interference with sleep.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
score on scale | 3.20 (0.17) | 2.44 (0.18) | 2.39 (0.17) | 2.26 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.76, 95% CI [-1.23 to -0.30]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.81, 95% CI [-1.27 to -0.34]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.94, 95% CI [-1.40 to -0.49]

13. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Sleep Disturbance
Description: Score range for sleep disturbance is 0-100.Higher scores indicate more of the attribute.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 86 | 93
score on scale | 31.99 (1.88) | 23.09 (2.00) | 23.75 (1.99) | 20.65 (1.88)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -8.90, 95% CI [-14.2 to -3.61]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.002, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -8.24, 95% CI [-13.5 to -2.99]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -11.3, 95% CI [-16.5 to -6.22]

14. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Snoring
Description: Score range for snoring is 0-100.Higher scores indicate more of the attribute.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 22.28 (2.57) | 26.58 (2.74) | 25.24 (2.73) | 31.99 (2.59)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.245, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 4.29, 95% CI [-2.95 to 11.54]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.417, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 2.95, 95% CI [-4.20 to 10.11]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.007, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 9.70, 95% CI [2.67 to 16.74]

15. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Awaken Short of Breath or With Headache
Description: Score range for awaken short of breath or with headache is 0-100. Higher scores indicate more of the attribute.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 5.99 (1.61) | 6.70 (1.72) | 6.70 (1.69) | 4.95 (1.62)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.760, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.71, 95% CI [-3.83 to 5.24]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.754, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.71, 95% CI [-3.75 to 5.18]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.641, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -1.04, 95% CI [-5.43 to 3.35]

16. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Quantity of Sleep
Description: Sleep Quantity subscale is scored from 0-24 indicating the number of hours of sleep. Higher scores indicate more of the attribute named in the subscale.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 6.58 (0.11) | 6.59 (0.12) | 6.85 (0.12) | 6.79 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.955, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.01, 95% CI [-0.30 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.084, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.27, 95% CI [-0.04 to 0.58]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.170, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.21, 95% CI [-0.09 to 0.52]

17. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Sleep Adequacy
Description: Score range for sleep adequacy is 0-100. Higher scores indicate more of the attribute.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 63.37 (2.67) | 67.38 (2.85) | 73.67 (2.82) | 69.37 (2.69)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.296, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 4.01, 95% CI [-3.52 to 11.55]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.007, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 10.30, 95% CI [2.87 to 17.73]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.106, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 6.00, 95% CI [-1.29 to 13.30]

18. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Somnolence
Description: Score range for Somnolence is 0-100. Higher scores indicate more of the attribute.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 30.23 (2.09) | 34.16 (2.23) | 41.45 (2.19) | 44.46 (2.10)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.191, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.93, 95% CI [-1.97 to 9.83]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 11.21, 95% CI [5.41 to 17.02]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 14.23, 95% CI [8.50 to 19.95]

19. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale Scores:Overall Sleep Problem Index
Description: Score range for overall sleep problem index is 0-100. Higher scores indicate more of the attribute.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 86 | 93
score on scale | 29.22 (1.50) | 25.19 (1.59) | 26.03 (1.58) | 26.78 (1.50)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.061, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -4.03, 95% CI [-8.25 to 0.18]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.133, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -3.20, 95% CI [-7.37 to 0.98]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.240, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -2.44, 95% CI [-6.52 to 1.64]

20. Secondary Outcome: Endpoint Medical Outcomes Study Sleep Scale: Number of Participants With Optimal Sleep
Description: Number of participants who reported Optimal Sleep
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
participants | 37 | 26 | 48 | 44
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.2842, Regression, Logistic; treatment, CLcr stratum, and the optimal sleep score at baseline as covariate; Odds Ratio (OR) = 0.68, 95% CI [0.34 to 1.37]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0577, Regression, Logistic; treatment, CLcr stratum, and the optimal sleep score at baseline as covariate; Odds Ratio (OR) = 1.89, 95% CI [0.98 to 3.66]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.1893, Regression, Logistic; treatment, CLcr stratum, and the optimal sleep score at baseline as covariate; Odds Ratio (OR) = 1.54, 95% CI [0.81 to 2.95]

21. Secondary Outcome: Endpoint Patient Global Impression Change
Description: Patient Global Impression Change is scaled from 1 to 7. 1=very much improved, 7=very much worse.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 3.6 (1.2) | 3.3 (1.2) | 2.9 (1.0) | 3.0 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0466, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; stratified by CLcr stratum

22. Secondary Outcome: Endpoint Clinical Global Impression Change
Description: Clinical Global Impression Change is scaled from 1 to 7. 1=very much improved, 7=very much worse.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 83 | 87 | 93
score on scale | 3.3 (1.1) | 3.1 (1.2) | 2.7 (1.1) | 2.7 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.3440, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; stratified by CLcr stratum
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; stratified by CLcr stratum

23. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Physical Functioning
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 76.16 (1.28) | 79.68 (1.37) | 76.93 (1.34) | 77.20 (1.28)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.057, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.51, 95% CI [-0.10 to 7.13]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.670, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.77, 95% CI [-2.78 to 4.32]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.559, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 1.04, 95% CI [-2.45 to 4.53]

24. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Role Limitations-Physical
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 67.96 (2.26) | 77.35 (2.41) | 74.63 (2.38) | 69.42 (2.28)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.004, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 9.40, 95% CI [3.01 to 15.78]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.037, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 6.67, 95% CI [0.39 to 12.95]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.643, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 1.46, 95% CI [-4.74 to 7.66]

25. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Bodily Pain
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 47.47 (1.82) | 48.09 (1.94) | 54.54 (1.91) | 52.50 (1.83)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.811, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 0.62, 95% CI [-4.50 to 5.75]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.006, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 7.07, 95% CI [2.03 to 12.12]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.047, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 5.03, 95% CI [0.06 to 10.00]

26. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: General Health Perception
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 52.36 (1.49) | 57.66 (1.59) | 56.19 (1.57) | 56.30 (1.50)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.013, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 5.30, 95% CI [1.10 to 9.50]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.070, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.82, 95% CI [-0.31 to 7.96]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.058, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.93, 95% CI [-0.13 to 8.00]

27. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Social Functioning
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 75.28 (2.20) | 77.71 (2.35) | 82.69 (2.32) | 77.11 (2.22)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.443, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 2.43, 95% CI [-3.79 to 8.65]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.018, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 7.41, 95% CI [1.28 to 13.54]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.549, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 1.83, 95% CI [-4.18 to 7.85]

28. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Role Limitations-Emotional
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 69.99 (2.40) | 76.14 (2.56) | 75.41 (2.52) | 73.02 (2.41)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.075, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 6.15, 95% CI [-0.63 to 12.92]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.111, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 5.41, 95% CI [-1.25 to 12.08]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.366, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.02, 95% CI [-3.55 to 9.60]

29. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Vitality
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 54.16 (1.90) | 59.80 (2.02) | 61.58 (2.00) | 58.31 (1.91)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.039, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 5.64, 95% CI [0.29 to 11.00]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.006, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 7.42, 95% CI [2.14 to 12.69]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.117, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 4.15, 95% CI [-1.05 to 9.34]

30. Secondary Outcome: Endpoint Short-Form 36-Item Health Survey Scores: Mental Health
Description: Short-Form 36-Item Health Survey is scored from 0-100 with higher scores reflecting better patient status.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
score on scale | 61.91 (1.95) | 65.90 (2.08) | 68.90 (2.05) | 66.67 (1.96)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.154, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 3.99, 95% CI [-1.50 to 9.49]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.012, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 6.99, 95% CI [1.58 to 12.40]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.079, ANCOVA; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = 4.76, 95% CI [-0.56 to 10.08]

31. Secondary Outcome: Number of Patients Not Reporting Allodynia
Description: Participants not reporting allodynia.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
participants | 65 | 52 | 63 | 66
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.6451, Regression, Logistic; treatment, CLcr stratum, and the presence of symptom at baseline as covariate; Odds Ratio (OR) = 1.28, 95% CI [0.45 to 3.59]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0745, Regression, Logistic; treatment, CLcr stratum, and the presence of symptom at baseline as covariate; Odds Ratio (OR) = 2.56, 95% CI [0.91 to 7.19]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.1787, Regression, Logistic; treatment, CLcr stratum, and the presence of symptom at baseline as covariate; Odds Ratio (OR) = 2.01, 95% CI [0.73 to 5.58]

32. Secondary Outcome: Number of Patients Not Reporting Hyperalgesia
Description: Participants not reporting hyperalgesia.
Time Frame: Week13/discontinuation
Population: Full analysis set. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 95 | 82 | 87 | 93
participants | 66 | 55 | 66 | 65
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0732, Regression, Logistic; treatment, CLcr stratum, and the presence of symptom at baseline as covariate; Odds Ratio (OR) = 2.26, 95% CI [0.93 to 5.52]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0353, Regression, Logistic; treatment, CLcr stratum, and the presence of symptom at baseline as covariate; Odds Ratio (OR) = 2.64, 95% CI [1.07 to 6.53]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.0393, Regression, Logistic; treatment, CLcr stratum, and the presence of symptom at baseline as covariate; Odds Ratio (OR) = 2.50, 95% CI [1.05 to 5.96]

33. Primary Outcome: Mean Pain Scores at Week 4
Description: as for outcome 4
Time Frame: Week4
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 92 | 82 | 78 | 82
score on scale | 5.43 (0.17) | 5.14 (0.18) | 4.57 (0.18) | 4.50 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.227, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.30, 95% CI [-0.78 to 0.18]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.86, 95% CI [-1.34 to -0.38]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.93, 95% CI [-1.40 to -0.46]

34. Primary Outcome: Mean Pain Scores at Week 5
Description: as for outcome 4
Time Frame: Week 5
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 90 | 81 | 77 | 78
score on scale | 5.29 (0.17) | 5.15 (0.18) | 4.42 (0.18) | 4.55 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.577, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.14, 95% CI [-0.62 to 0.35]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Median Difference (Final Values) = -0.87, 95% CI [-1.35 to -0.39]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.002, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.74, 95% CI [-1.22 to -0.27]

35. Primary Outcome: Mean Pain Scores at Week 6
Description: as for outcome 4
Time Frame: Week 6
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 89 | 80 | 77 | 78
score on scale | 5.29 (0.17) | 5.02 (0.18) | 4.31 (0.18) | 4.54 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.275, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.27, 95% CI [-0.75 to 0.21]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.98, 95% CI [-1.46 to -0.50]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.002, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.75, 95% CI [-1.22 to -0.28]

36. Primary Outcome: Mean Pain Scores at Week 7
Description: as for outcome 4
Time Frame: Week 7
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 88 | 80 | 75 | 78
score on scale | 5.14 (0.17) | 4.90 (0.18) | 4.24 (0.18) | 4.48 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.334, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.24, 95% CI [-0.72 to 0.25]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.90, 95% CI [-1.38 to -0.42]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.006, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.66, 95% CI [-1.14 to -0.19]

37. Primary Outcome: Mean Pain Scores at Week 8
Description: as for outcome 4
Time Frame: Week 8
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 88 | 79 | 75 | 76
score on scale | 5.04 (0.17) | 4.89 (0.18) | 4.23 (0.18) | 4.47 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.530, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.15, 95% CI [-0.64 to 0.33]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.82, 95% CI [-1.30 to -0.33]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.017, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.58, 95% CI [-1.05 to -0.10]

38. Primary Outcome: Mean Pain Scores at Week 9
Description: as for outcome 4
Time Frame: Week 9
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 86 | 78 | 73 | 74
score on scale | 5.08 (0.17) | 4.87 (0.18) | 4.22 (0.18) | 4.50 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.392, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.21, 95% CI [-0.70 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.87, 95% CI [-1.35 to -0.38]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.016, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.58, 95% CI [-1.06 to -0.11]

39. Primary Outcome: Mean Pain Scores at Week 10
Description: as for outcome 4
Time Frame: Week 10
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 86 | 77 | 72 | 72
score on scale | 5.08 (0.17) | 4.86 (0.18) | 4.18 (0.18) | 4.56 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.364, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.22, 95% CI [-0.71 to 0.26]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.91, 95% CI [-1.39 to -0.42]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.031, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.52, 95% CI [-1.00 to -0.05]

40. Primary Outcome: Mean Pain Scores at Week 11
Description: as for outcome 4
Time Frame: Week 11
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 85 | 75 | 72 | 71
score on scale | 5.12 (0.17) | 4.88 (0.18) | 4.18 (0.18) | 4.47 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.326, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.24, 95% CI [-0.73 to 0.24]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p < 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.94, 95% CI [-1.43 to -0.46]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.007, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.65, 95% CI [-1.13 to -0.18]

41. Primary Outcome: Mean Pain Scores at Week 12
Description: as for outcome 4
Time Frame: Week 12
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 83 | 74 | 72 | 71
score on scale | 5.00 (0.17) | 4.71 (0.18) | 4.15 (0.18) | 4.37 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.241, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.29, 95% CI [-0.78 to 0.20]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.85, 95% CI [-1.34 to -0.37]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.010, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.63, 95% CI [-1.10 to -0.15]

42. Primary Outcome: Mean Pain Scores at Week 13
Description: as for outcome 4
Time Frame: Week 13
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 82 | 73 | 72 | 71
score on scale | 4.97 (0.17) | 4.70 (0.18) | 4.16 (0.18) | 4.36 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.281, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.27, 95% CI [-0.76 to 0.22]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 300 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.001, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.82, 95% CI [-1.30 to -0.33]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 600 mg/Day; Hypothesis testing was conducted using two-sided tests with significance level of 0.05; Test type: Superiority or Other; p = 0.012, repeated measures analysis; The model included treatment and CLcr stratum as factors, and baseline score as covariate; Mean Difference (Final Values) = -0.62, 95% CI [-1.09 to -0.14]

43. Secondary Outcome: Mean Sleep Interference Scores at Week 1
Description: Weekly mean sleep interference scores is defined as the mean of the last 7 daily diary interference with sleep ratings. Scores range from 0-10 (11 points ordinal) with higher scores indicating more severe interference with sleep.
Time Frame: week 1
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 97 | 86 | 89 | 97
score on scale | 3.79 (0.15) | 3.00 (0.16) | 2.97 (0.16) | 2.81 (0.15)

44. Secondary Outcome: Mean Sleep Interference Scores at Week 2
Description: as for outcome 43
Time Frame: week 2
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 96 | 83 | 83 | 86
score on scale | 3.56 (0.15) | 2.89 (0.16) | 2.76 (0.16) | 2.49 (0.15)

45. Secondary Outcome: Mean Sleep Interference Scores at Week 3
Description: as for outcome 43
Time Frame: week 3
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 92 | 83 | 80 | 84
score on scale | 3.50 (0.15) | 2.81 (0.16) | 2.60 (0.16) | 2.43 (0.15)

46. Secondary Outcome: Mean Sleep Interference Scores at Week 4
Description: as for outcome 43
Time Frame: week 4
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 92 | 82 | 78 | 82
score on scale | 3.35 (0.15) | 2.79 (0.16) | 2.54 (0.16) | 2.36 (0.15)

47. Secondary Outcome: Mean Sleep Interference Scores at Week 5
Description: as for outcome 43
Time Frame: week 5
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 90 | 81 | 77 | 78
score on scale | 3.26 (0.15) | 2.74 (0.16) | 2.39 (0.16) | 2.41 (0.15)

48. Secondary Outcome: Mean Sleep Interference Scores at Week 6
Description: as for outcome 43
Time Frame: week 6
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 89 | 80 | 77 | 78
score on scale | 3.24 (0.15) | 2.63 (0.16) | 2.37 (0.16) | 2.33 (0.15)

49. Secondary Outcome: Mean Sleep Interference Scores at Week 7
Description: as for outcome 43
Time Frame: week 7
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 88 | 80 | 75 | 78
score on scale | 3.19 (0.15) | 2.55 (0.16) | 2.36 (0.16) | 2.21 (0.15)

50. Secondary Outcome: Mean Sleep Interference Scores at Week 8
Description: as for outcome 43
Time Frame: week 8
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 88 | 79 | 75 | 76
score on scale | 3.10 (0.15) | 2.49 (0.16) | 2.30 (0.16) | 2.14 (0.15)

51. Secondary Outcome: Mean Sleep Interference Scores at Week 9
Description: as for outcome 43
Time Frame: week 9
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 86 | 78 | 73 | 74
score on scale | 3.17 (0.15) | 2.44 (0.16) | 2.38 (0.16) | 2.22 (0.16)

52. Secondary Outcome: Mean Sleep Interference Scores at Week 10
Description: as for outcome 43
Time Frame: week 10
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 86 | 77 | 72 | 72
score on scale | 3.16 (0.15) | 2.46 (0.16) | 2.39 (0.16) | 2.28 (0.16)

53. Secondary Outcome: Mean Sleep Interference Scores at Week 11
Description: as for outcome 43
Time Frame: week 11
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 85 | 75 | 72 | 71
score on scale | 3.16 (0.15) | 2.43 (0.16) | 2.37 (0.16) | 2.27 (0.16)

54. Secondary Outcome: Mean Sleep Interference Scores at Week 12
Description: as for outcome 43
Time Frame: week 12
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 83 | 74 | 72 | 71
score on scale | 3.06 (0.15) | 2.36 (0.16) | 2.28 (0.16) | 2.21 (0.16)

55. Secondary Outcome: Mean Sleep Interference Scores at Week 13
Description: as for outcome 43
Time Frame: week 13
Population: Full analysis set. Observed case.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 82 | 73 | 72 | 71
score on scale | 3.08 (0.15) | 2.33 (0.16) | 2.27 (0.16) | 2.19 (0.16)

ADVERSE EVENTS:
Arm/Group | Placebo | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 600 mg/Day
Serious Adverse Events (participants affected / at risk) | 6/98 | 2/87 | 4/89 | 1/97
Other Adverse Events (participants affected / at risk) | 35/98 | 44/87 | 61/89 | 77/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=98) | Pregabalin 150 mg/Day (N=87) | Pregabalin 300 mg/Day (N=89) | Pregabalin 600 mg/Day (N=97)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Large intestinal stricture (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=98) | Pregabalin 150 mg/Day (N=87) | Pregabalin 300 mg/Day (N=89) | Pregabalin 600 mg/Day (N=97)
Diplopia (Eye disorders) | 0 | 0 | 2 | 6
Constipation (Gastrointestinal disorders) | 6 | 12 | 11 | 14
Nausea (Gastrointestinal disorders) | 5 | 2 | 6 | 7
Face oedema (General disorders) | 0 | 4 | 1 | 6
Oedema peripheral (General disorders) | 1 | 4 | 12 | 18
Thirst (General disorders) | 3 | 3 | 7 | 7
Nasopharyngitis (Infections and infestations) | 10 | 8 | 10 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 5 | 4 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 7 | 4
Weight increased (Investigations) | 0 | 1 | 17 | 14
Dizziness (Nervous system disorders) | 7 | 10 | 27 | 48
Headache (Nervous system disorders) | 1 | 2 | 1 | 5
Somnolence (Nervous system disorders) | 9 | 19 | 22 | 37
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.